CLINICAL TRIAL: NCT07196644
Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Telisotuzumab Adizutecan for the Treatment of Subjects With Locally Advanced or Metastatic Solid Tumors That Harbor MET Amplification
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity in Participants 12 Years of Age or Older With Locally Advanced or Metastatic Solid Tumors That Harbor MET Amplification Receiving Intravenously Infused Telisotuzumab Adizutecan
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M25-279; 2024-518871-74 (Other: EU CT)
Record Dates: First submitted 2025-09-22; First posted 2025-09-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Solid Tumors Harboring MET Amplification
Keywords: Solid Tumors harboring MET Amplification; Telisotuzumab Adizutecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Telisotuzumab Adizutecan (Experimental): Participants will receive telisotuzumab adizutecan, as part of the 61.5 month study duration.
  Interventions: Drug: Telisotuzumab Adizutecan

INTERVENTIONS:
Drug: Telisotuzumab Adizutecan — Intravenous (IV) Infusion

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. The purpose of this study is to assess adverse events and change in disease activity of telisotuzumab adizutecan.

Telisotuzumab adizutecan is an investigational drug being developed for the treatment of locally advanced or metastatic solid tumors that harbor MET amplification. This study will have 1 arm where participants will receive telisotuzumab adizutecan. Approximately 125 participants 12 years of age or older. with solid tumors harboring MET amplification will be enrolled in the study in up to 55 sites around the world.

Participants will receive intravenous (IV) telisotuzumab adizutecan, as part of the 61.5 month study duration.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced/metastatic solid tumors with documented MET amplification via Local next generation sequencing (NGS) or Central NGS via FoundationOne Companion Diagnostic (F1CDx).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1
* Measurable disease at baseline per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 or Response Assessment in Neuro-Oncology (RANO) criteria as appropriate to tumor type.
* Received prior systemic therapy appropriate for their tumor type and stage of disease and who have no satisfactory alternative therapy for advanced solid tumors that would be expected to provide a substantial survival benefit for their tumor type.
* If participant has central nervous system (CNS) metastasis, these should be clinically asymptomatic or radiologically stable (i.e., without evidence of progression after definitive treatment

Exclusion Criteria:

* Current, historical, or suspected (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids.
* Any major, life-threatening conditions and life expectancy should be at least 12 weeks.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-10-29 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events (AE)s | Up to 61.5 Months
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.
Confirmed Objective Response (OR) as Assessed by Independent Central Review (ICR) | Up to 36 Months
  OR is defined as (subjects achieving complete response [CR] or partial response [PR]) as assessed by ICR based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or Response Assessment in Neuro-Oncology (criteria) (RANO) criteria as appropriate to tumor type in participants with MET amplified positivity determined by FoundationOne CDx (F1CDx) testing.

SECONDARY OUTCOMES:
Duration of Response (DoR) as Assessed by ICR in participants with MET amplified positivity determined by F1CDx testing | Up to 36 Months
  DoR is defined for confirmed responders as the time from the first documented response (initial CR or PR) until the first occurrence of radiographic progression per ICR based on RECIST v1.1 or RANO criteria as appropriate to tumor type or death from any cause, whichever occurs first.
Progression-Free Survival (PFS) as Assessed by ICR in participants with MET amplified positivity determined by F1CDx testing | Up to 36 Months
  DoR is defined for confirmed responders as the time from the first documented response (initial CR or PR) until the first occurrence of radiographic progression per ICR based on RECIST v1.1 or RANO criteria as appropriate to tumor type or death from any cause, whichever occurs first.
Disease Control (DC) as Assessed by ICR based on RECIST v1.1 or RANO criteria as appropriate to tumor type in subjects with MET amplified positivity determined by F1CDx testing | Up to 36 Months
  DC is defined as achieving an OR or stable disease (SD) according to RECIST v1.1 by investigator at any time prior to subsequent anti-cancer therapy.
OS in Participants with MET Amplified Positivity Determined by F1CDx Testing | Up to 36 Months
  OS is defined as the time from first dose until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- United States (8):
  - Valkyrie Clinical Trials /ID# 275547, Los Angeles, California
  - Northwestern University Feinberg School of Medicine /ID# 276436, Chicago, Illinois
  - University of Chicago Medical Center /ID# 275342, Chicago, Illinois
  - START Midwest /ID# 276603, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center - New York - York Avenue /ID# 275999, New York, New York
  - Duke Cancer Institute /ID# 275604, Durham, North Carolina
  - South Texas Accelerated Research Therapeutics (START) /ID# 276608, San Antonio, Texas
  - Start Mountain Region /ID# 276607, West Valley City, Utah
- Israel (4):
  - The Chaim Sheba Medical Center /ID# 274342, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 274344, Tel Aviv, Tel Aviv
  - Hadassah Medical Center-Hebrew University /ID# 274343, Jerusalem
  - Rabin Medical Center. /ID# 274341, Petah Tikva
- Japan (6):
  - Nagoya University Hospital /ID# 276336, Nagoya, Aichi-ken
  - Hokkaido University Hospital /ID# 276333, Sapporo, Hokkaido
  - Kyoto University Hospital /ID# 276398, Kyoto, Kyoto
  - Tohoku University Hospital /ID# 276344, Sendai, Miyagi
  - Okayama University Hospital /ID# 276299, Okayama, Okayama-ken
  - National Cancer Center Hospital /ID# 276297, Chuo-Ku, Tokyo
- South Korea (3):
  - Seoul National University Hospital /ID# 275703, Seoul, Seoul Teugbyeolsi
  - Yonsei University Health System Severance Hospital /ID# 276184, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 275705, Seoul, Seoul Teugbyeolsi

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-279